CLINICAL TRIAL: NCT03987620
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Oral Ibrexafungerp (SCY-078) vs. Placebo in Subjects With Acute Vulvovaginal Candidiasis (AVVC).
Brief Title: Efficacy and Safety of Oral Ibrexafungerp (SCY-078) vs. Placebo in Subjects With Acute Vulvovaginal Candidiasis
Acronym: Vanish 306
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCY-078-306
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Candida Vulvovaginitis
Keywords: Vaginitis; Yeast infection
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Vaginitis | interventions — ibrexafungerp

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibrexafungerp (SCY-078) (Experimental): 300 mg BID for one day
  Interventions: Drug: Ibrexafungerp
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibrexafungerp — Ibrexafungerp 300mg BID for one day
  Other Names: SCY-078
  Arms: Ibrexafungerp (SCY-078)
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, multicenter, double-blind, placebo-controlled study to evaluate the efficacy and safety of oral Ibrexafungerp (SCY-078) compared to placebo in female subjects 12 years and older with AVVC.

DETAILED DESCRIPTION:
Subjects who meet all of the inclusion and none of the exclusion criteria will be enrolled into the study and will be randomized in a 2:1 ratio to either oral ibrexafungerp or ibrexafungerp matching placebo, as follows:

* Oral ibrexafungerp 300-mg dose BID (bis in die) for 1 day
* Oral ibrexafungerp matching placebo BID for 1 day

This is a randomized, double-blind study.

Approximately 366 eligible subjects will be enrolled and randomized in a 2:1 ratio to one of the two study treatment groups. Subjects will be followed for assessments of efficacy and safety for approximately one month after study drug administration. The design of this study is identical to VANISH 303 Study: NCT03734991

ELIGIBILITY:
Inclusion Criteria:

* Subject is a postmenarchal female subject 12 years and older
* Subject has a diagnosis of symptomatic AVVC at baseline including a positive microscopic examination with 10% Potassium Hydroxide (KOH) in a vaginal sample revealing yeast forms (hyphae/pseudohyphae) or budding yeasts, and vaginal pH (≤4.5)

Exclusion Criteria:

* Subject has any vaginal condition other than AVVC that may interfere with the diagnosis or evaluation of response to therapy, such as suspected or confirmed concurrent causes of vulvovaginitis and/or cervicitis (mixed infection)
* Need for systemic and/or topical (vaginal) anti fungal treatment, including prescription or over-the-counter products during the study and treatment for vulvovaginal candidiasis (VVC) 28 days prior to randomization.
* Subject has uncontrolled diabetes mellitus.
* Subject has a vaginal sample with pH >4.5.
* Subject has a history of or an active cervical/vaginal cancer.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 455 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2020-04-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (21):
  - Mesa OB-GYN, Mesa, Arizona
  - Red Rocks OBGYN, Lakewood, Colorado
  - Planned Parenthood Southern New England, New Haven, Connecticut
  - New Generation Medical Research, Hialeah, Florida
  - Healthcare Clinical Data Inc, North Miami, Florida
  - Physician Care Clinical Research LLC, Sarasota, Florida
  - CCT LLC - A VitaLink Company- PPDS, West Palm Beach, Florida
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Fellows Research Alliance Inc, Savannah, Georgia
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Praetorian Pharmaceutical Research, LLC, Marrero, Louisiana
  - North County Health Center, Planned Parenthood of the St. Louis Region and Southwest Missouri, Florissant, Missouri
  - Clinical Research Center Of Nevada, Las Vegas, Nevada
  - Planned Parenthood North Central Southern New Jersey (PPNCSNJ), Hackensack, New Jersey
  - Carolina Institute for Clinical Research - M3 Wake Research, Fayetteville, North Carolina
  - Obstetrics and Gynecology Associates of Erie, PC, Erie, Pennsylvania
  - Planned Parenthood Southeastern Pennsylvania The Elizabeth Blackwell Health Center, Philadelphia, Pennsylvania
  - Fellows Research Alliance Inc, Bluffton, South Carolina
  - Chattanooga Medical Research Inc, Chattanooga, Tennessee
  - Signature GYN Services, PLLC, Fort Worth, Texas
  - Brownstone Clinical Trials, LLC, Irving, Texas
- Bulgaria (20):
  - Multiprofile Hospital for Active Treatment -Asenovgrad EOOD, Asenovgrad
  - MHAT Puls AD - PPDS, Blagoevgrad
  - Multiprofile Hospital for Active Treatment - Chirpan EOOD, Chirpan
  - Medical Center Asklepii OOD, Dupnitsa
  - Diagnostic-Consultative Center I-Gabrovo EOOD, Gabrovo
  - Multiprofile Hospital For Active Treatment Dr Tota Venkova, Gabrovo
  - Multiprofile Hospital for Active Treatment Sv. Ivan Rilski - Gorna Oryahovitsa EOOD, Gorna Oryahovitsa
  - Multiprofile Hospital for Active Treatment- Sveti Nikolay Chudotvoretz - LOM EOOD, Lom
  - Multiprofile Hospital for Active Treatment - Prof. Dr. Paraskev Stoyanov AD, Lovech
  - MHAT Stamen Iliev AD, Montana
  - Multiprofile Hospital For Active Treatment - Pazardzhik AD, Pazardzhik
  - Multiprofile Hospital for Active Treatment Trimontsium OOD, Plovdiv
  - Multiprofile Hospital for Active Treatment - Samokov EOOD, Samokov
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - Multiprofile Hospital for Active Treatment Shumen, Shumen
  - Multiprofile Hospital For Active Treatment - Dr. Bratan Shukerov AD, Smolyan
  - Medical Center Excelsior OOD - PPDS, Sofia
  - Diagnostic Consultative CTR - XX - Sofia - EOOD, Sofia
  - Medical center Vip Clinic OOD, Sofia
  - Medical Center Medica Plus OOD, Veliko Tarnovo

REFERENCES:
- [Derived] Goje O, Sobel R, Nyirjesy P, Goldstein SR, Spitzer M, Faught B, Larson S, King T, Azie NE, Angulo D, Sobel JD. Oral Ibrexafungerp for Vulvovaginal Candidiasis Treatment: An Analysis of VANISH 303 and VANISH 306. J Womens Health (Larchmt). 2023 Feb;32(2):178-186. doi: 10.1089/jwh.2022.0132. Epub 2022 Oct 17. PMID 36255448

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 22 medical center between 07Jun2019 and 07Feb2020.
Period: Overall Study
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Started | 303 | 152
Withdrawn Before Treatment | 5 | 1
Withdrawn Before TOC | 48 | 45
Completed the TOC Visit | 250 | 106
Withdrawn At or After the TOC Visit | 4 | 4
Completed | 246 | 102
Not Completed | 57 | 50
Not completed — Lack of Efficacy or Use of antifungal therapy | 43 | 41
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Other | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrexafungerp (SCY-078) | Placebo | Total
Number analyzed (Participants) | 298 | 151 | 449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 296 | 149 | 445
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (10.45) | 34.5 (10.94) | 34.2 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 151 | 449
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 14 | 50
  Not Hispanic or Latino | 262 | 137 | 399
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 51 | 27 | 78
  White | 246 | 123 | 369
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 105 | 66 | 171
  Bulgaria | 193 | 85 | 278

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure (Complete Resolution of Signs and Symptoms)
Description: The percentage of subjects with clinical cure (complete resolution of signs and symptoms) at the test-of-cure (TOC) visit
Time Frame: Day 8-14
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Number analyzed (Participants) | 188 | 84
Participants
  Clinical cure | 119 | 37
  Clinical failure | 69 | 47

2. Secondary Outcome: Mycological Eradication (Negative Culture for Growth of Yeast)
Description: The percentage of subjects with mycological eradication (negative culture for growth of Candida species) at the TOC visit
Time Frame: Day 8-14
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Number analyzed (Participants) | 188 | 84
Participants
  Mycological eradication | 110 | 25
  Mycological persistence | 78 | 59

3. Secondary Outcome: Clinical Cure and Mycological Eradication (Responder Outcome)
Description: The percentage of subjects with clinical cure and mycological eradication (responder outcome) at the TOC visit
Time Frame: Day 8-14
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Number analyzed (Participants) | 178 | 81
Participants
  Overall success | 82 | 23
  Overall failure | 96 | 58

4. Secondary Outcome: Complete Clinical Response at Follow-up
Description: The percentage of subjects with complete resolution of signs and symptoms at the Follow-up (FU) visit
Time Frame: Day 25
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Number analyzed (Participants) | 189 | 89
Participants
  Clinical cure at Follow up | 137 | 44
  Clinical failure at Follow up | 52 | 45

5. Secondary Outcome: Safety and Tolerability of Ibrexafungerp
Description: Number of subjects with treatment related adverse events
Time Frame: Up to 29 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Number analyzed (Participants) | 100 | 45
Participants
  Any treatment-emergent adverse event | 99 | 44
  Any serious treatment-emergent adverse event | 1 | 1
  Any treatment-related treatment-emergent serious adverse event | 0 | 0
  Any treatment-emergent adverse event leading to treatment discontinuation | 0 | 0
  Any adverse event leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks after last dose
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/298 | 0/151
Serious Adverse Events (participants affected / at risk) | 1/298 | 1/151
Other Adverse Events (participants affected / at risk) | 63/298 | 15/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp (SCY-078) (N=298) | Placebo (N=151)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Gastrointestinal bacterial infection (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp (SCY-078) (N=298) | Placebo (N=151)
Diarrhoea (Gastrointestinal disorders) | 28 | 1
Nausea (Gastrointestinal disorders) | 25 | 4
Headache (Nervous system disorders) | 22 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT03987620/Prot_001.pdf
  • Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT03987620/SAP_002.pdf